CLINICAL TRIAL: NCT02218424
Title: Systemic Magnesium to Improve Postoperative Pain in Pediatric Patients Undergoing Tonsillectomy: A Randomized, Double Blinded, Placebo Controlled Trial
Brief Title: Magnesium vs Placebo for Tonsillectomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Hubert Benzon, Principal Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014MagRCT
Record Dates: First submitted 2014-08-12; First posted 2014-08-18 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Magnesium; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium (Experimental): Intravenous magnesium. After IV placed intraoperatively, a bolus dose of magnesium 30 mg/kg is given over 15 minutes, followed by a continuous infusion of magnesium at 10 mg/kg/hr until the completion of the procedure.
  Interventions: Drug: Magnesium
- Placebo infusion (Placebo Comparator): Intravenous normal saline will be given as placebo. An equal amount of volume normal saline will be given intravenously as the control group.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Magnesium
  Arms: Magnesium
Drug: Normal saline
  Arms: Placebo infusion

SUMMARY:
This study is a double-blind randomized controlled trial using intravenous magnesium versus placebo to determine if systemic magnesium can decrease postoperative pain in pediatric patients undergoing tonsillectomy.

Participants will be in one of two arms. Those in Arm 1 will receive magnesium (30 mg/kg bolus followed by a 10mg/kg/hr infusion) while those in Arm 2 will receive an equal volume of normal saline bolus followed by infusion (placebo).

The primary objective is to determine if systemic magnesium will decrease postoperative pain in patients undergoing tonsillectomy. The secondary objectives will determine if systemic magnesium administration is associated with a decrease in opioid-related side effects, decrease the incidence of emergence delirium, and improve postoperative functional recovery.

The study hypothesis is that the use of intravenous magnesium will decrease postoperative pain, decrease opioid-related side effects, decrease the incidence of emergence delirium, and improve functional recovery in patients undergoing tonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 4-10 years old undergoing tonsillectomy by a single surgeon and under the care of that participating surgeon
* American Society of Anesthesiology (ASA) patient classification of I-III

Exclusion Criteria:

* Physical or developmental delay
* Psychiatric illness
* Current use of sedative or anticonvulsant medication
* Pre-existing renal disease
* Pre-existing cardiovascular disease
* Regular use of analgesic medication
* Having other procedures in addition to tonsillectomy (however, patients undergoing adenoidectomy with their tonsillectomy will be included in the study)

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hubert A Benzon, MD, MPH, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Magnesium: Intravenous magnesium. After IV placed intraoperatively, a bolus dose of magnesium 30 mg/kg is given over 15 minutes, followed by a continuous infusion of magnesium at 10 mg/kg/hr until the completion of the procedure.
  Magnesium
- Placebo Infusion: Intravenous normal saline will be given as placebo. An equal amount of volume normal saline will be given intravenously as the control group.
  Normal saline
Period: Overall Study
Arm/Group | Magnesium | Placebo Infusion
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium | Placebo Infusion | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: Months] | 76.5 [65 to 94] | 76.5 [61 to 92] | 76.5 [63 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m2] | 16.1 [14.3 to 18.2] | 16.9 [14.4 to 20.0] | 16.4 [14.2 to 19.8]
Obstructive Sleep Apnea (Yes/No) [Count of Participants; unit: Participants]
  Yes | 7 | 8 | 15
  No | 23 | 22 | 45
Surgical Duration [Median (Inter-Quartile Range); unit: Minutes] | 36.5 [32 to 40] | 35 [33 to 39] | 35 [33 to 40]

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain
Description: Postoperative pain will be measured at 15 minute time intervals in the post-anesthesia care unit (PACU). Pain scores will be evaluated using a standardized validated scale (the Faces Pain Scale Revised (FPS-R)). The Faces Pain Scale is a validated, patient reported, 0 (no pain) to 10 (worst pain imaginable) numeric rating scale. Pain scores will be multiplied by the time spent at each pain score for a calculated "Area Under the Curve" value, ranging from 0 to 900, with lower values indicating more favorable and lower pain scores.
Time Frame: 90 minutes
Measure: Median (Inter-Quartile Range); unit: scores on a scale*minutes
Arm/Group | Magnesium | Placebo Infusion
Number analyzed (Participants) | 30 | 30
scores on a scale*minutes | 30 [0 to 120] | 45 [0 to 135]

2. Secondary Outcome: Postoperative Pain Medication
Description: Amount of rescue postoperative pain medication needed in the recovery room will be tabulated.
Time Frame: 90 minutes
Measure: Median (Inter-Quartile Range); unit: mg IV morphine
Arm/Group | Magnesium | Placebo Infusion
Number analyzed (Participants) | 30 | 30
mg IV morphine | 2.0 [0.0 to 4.44] | 2.5 [0 to 4.99]

3. Secondary Outcome: Postoperative Pain at Home
Description: Postoperative pain at home will be measured using the Parent's Post-Operative Pain Measure (PPPM) questionnaire on postoperative days 1, 3, and 7. The PPPM gives a score to child behavior which suggests they are in pain after surgery with scores ranging from 0 to 15 with lower values suggesting better pain outcome.
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: PPPM Scale Score (Range: 0-15)
Arm/Group | Magnesium | Placebo Infusion
Number analyzed (Participants) | 30 | 30
PPPM Scale Score (Range: 0-15) | 5.5 [4 to 7] | 5 [2 to 7]

4. Secondary Outcome: Emergence Delirium
Description: The incidence of emergence delirium determined using the pediatric anesthesia emergence delirium (PAED) scale while the patient is in the PACU. The PAED scale ranges from scores of 0 to 20, with lower scores indicating less agitation, more awareness, less aggressiveness, and a more favorable outcome in the post-anesthesia recovery period.
Time Frame: 5 minutes after awakening in the recovery room
Measure: Median (Inter-Quartile Range); unit: Units on a scale, PAED
Arm/Group | Magnesium | Placebo Infusion
Number analyzed (Participants) | 30 | 30
Units on a scale, PAED | 5 [3 to 11] | 6.5 [0 to 12]

5. Secondary Outcome: Number of Patients With Postoperative Vomiting
Description: The incidence of postoperative vomiting will be measured while in the recovery room.
Time Frame: 90 minutes
Measure: Number; unit: participants
Arm/Group | Magnesium | Placebo Infusion
Number analyzed (Participants) | 30 | 30
participants | 0 | 0

6. Secondary Outcome: Respiratory Depression
Description: The incidence of the presence of respiratory depression will be measured while the patient is in the recovery room.
Time Frame: 90 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Magnesium | Placebo Infusion
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

7. Secondary Outcome: Time to PACU Discharge
Description: The time to fulfilling discharge criteria, in minutes, from the PACU will be recorded
Time Frame: Approximately 90 minutes
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Magnesium | Placebo Infusion
Number analyzed (Participants) | 30 | 30
Minutes | 57 (19) | 62 (16)

8. Secondary Outcome: Parent Satisfaction
Description: Parent satisfaction will be assessed on postoperative days 1, 3, and 7. This will be determined by asking the parents one question about their satisfaction with the overal anesthetic care on a numeric rating scale of 1 to 10, with higher scores indicating greater satisfaction and better outcome.
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: Units on a Numeric Rating Scale
Arm/Group | Magnesium | Placebo Infusion
Number analyzed (Participants) | 30 | 30
Units on a Numeric Rating Scale | 10 [10 to 10] | 10 [10 to 10]

ADVERSE EVENTS:
Arm/Group | Magnesium | Placebo Infusion
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No